CLINICAL TRIAL: NCT01730352
Title: Helicobacter Pylori Infection and Chronic Immune Thrombocytopenic Purpura in Children and Adolescents - A Randomized Controlled Trial
Brief Title: Helicobacter Pylori Treatment in Immune Thrombocytopenic Purpura (ITP) Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Elisabete Kawakami, Professor, PhD MD, Federal University of São Paulo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 08/56706-0
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Immune Thrombocytopenic Purpura; Helicobacter Pylori Infection
Keywords: immune thrombocytopenic purpura; chronic immune thrombocytopenic purpura; secondary immune thrombocytopenic purpura; Helicobacter pylori infection; Helicobacter pylori gastritis; children; adolescents
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- H. pylori no treatment (No Intervention): Observational group, with clinical and platelet count follow-up
- H. pylori triple therapy (Experimental): Triple therapy for H. pylori eradication: clarithromycin 15mg/kg, amoxicillin 50mg/kg, furazolidone 7mg/kg and/ or doxycycline 4,4mg/kg (all 2 times per day), with a proton pump inhibitor for 14 days.
  Interventions: Drug: H. pylori triple therapy

INTERVENTIONS:
Drug: H. pylori triple therapy — Children up to 5 years: clarithromycin 15mg/kg, amoxicillin 50mg/kg, and/or furazolidone 7mg/kg Children above 8 years: doxycycline 4,4mg/kg if necessary Children able to swallow tablets or capsules, above 30kg: clarithromycin 500mg, amoxicillin 500mg, furazolidone 200mg, and/ or doxycycline 100mg, all 2 times per day, for 14 days.
  Other Names: Triple therapy for H. pylori; H. pylori eradication therapy; Pyloripac
  Arms: H. pylori triple therapy

SUMMARY:
The purpose of this study is to determine whether eradication of Helicobacter pylori infection is effective in the improvement of platelet counts in children and adolescents with chronic ITP.

DETAILED DESCRIPTION:
Helicobacter pylori infection has been associated with Immune Thrombocytopenic Purpura (ITP), and there is scientific evidence for the investigation and treatment of this bacterium for adult patients with ITP. However, in children this causal association is not clear, with few published studies.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of chronic immune thrombocytopenic purpura
* children and adolescents up to 20 years

Exclusion Criteria:

* known hypersensitivity to any of the drugs
* recent treatment for H. pylori eradication

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2008-10; Primary Completion 2011-05 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
platelet response | 1 year
  Responders: Complete Response (CR), persistent elevation of platelet count to >150×109/L; Partial Response (PR), elevation between 20 and 30×109/L above the baseline values, but between 50 and 149×109/L; No Responders: any of the above categories.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabete Kawakami, Professor, Principal Investigator — Federal University of São Paulo
Locations (4):
- Brazil (4):
  - Irmandade da Santa Casa de Misericordia se Sao Paulo, São Paulo, São Paulo
  - Centro de Hematologia de Sao Paulo, São Paulo, São Paulo
  - Federal University of Sao Paulo, São Paulo, São Paulo
  - Hospital Estadual Infantil Darcy Vargas, São Paulo, São Paulo